CLINICAL TRIAL: NCT00270517
Title: A Randomized, Double-Blinded, Parallel Group, Multicenter Study of EDP-420 Versus Telithromycin for the Treatment of Community Acquired Pneumonia
Brief Title: Comparative Study of EDP-420 Versus Another Antibiotic in the Treatment of Community Acquired Pneumonia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDP420-05-006
Record Dates: First submitted 2005-12-23; First posted 2005-12-28 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2006-09

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — EDP 420; Duration of Therapy; telithromycin

INTERVENTIONS:
Drug: EDP-420 / Duration of Treatment - 3 days
Drug: Telithromycin / Duration of Treatment - 7 days

SUMMARY:
This study will compare the efficacy, safety and tolerability of EDP-420 versus another oral antibiotic in the treatment of community acquired pneumonia

ELIGIBILITY:
Inclusion Criteria:

* Recent respiratory illness with signs and symptoms and chest X-ray consistent with the diagnosis of community-acquired pneumonia.
* Suitable candidate for oral antibiotic therapy and able to swallow large capsules intact
* If female, must be non-lactating and at no risk for pregnancy

Exclusion Criteria:

* Other infections
* Other pulmonary diseases requirement multiple antibacterial medications or long duration of therapy
* History of hypersensitivity, allergic or adverse reactions to macrolide, ketolide, azalide or streptogramins
* Evidence of uncontrolled clinically significant disease, malignancy, or other abnormality
* Requirement of parenteral antimicrobial therapy for treatment of pneumonia
* Currently receiving or likely to receive any known inhibitors or inducers of cytochrome P450 mediated drug metabolism
* Immunocompromised subjects

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2005-12; Study Completion 2007-07

PRIMARY OUTCOMES:
Clinical Cure 7-14 days after end of therapy

SECONDARY OUTCOMES:
Bacteriological response
Radiographic response
Change in signs and symptoms
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- Enanta Pharmaceuticals, Inc., Watertown, Massachusetts, United States